CLINICAL TRIAL: NCT01070160
Title: Endometrial Effects of Metformin Action in Women With Polycystic Ovarian Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0905005203; U54HD052668-02 (NIH)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2014-06

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: Polycystic Ovarian Syndrome (PCOS); Metformin; Endometrin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Progesterone; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, endometrium tissue biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Women with PCOS initiating Metformin and exposure to vaginal progesterone for 6-8 days prior ro Endometrium Biopsy
  Interventions: Drug: Endometrin (progesterone 100mg vaginal inserts); Drug: Metformin
- B: Women with PCOS not planning initiating Metformin and exposure to vaginal progesterone for 6-8 days prior to Endometrium Biopsy
  Interventions: Drug: Endometrin (progesterone 100mg vaginal inserts)
- Women with PCOS who previously initiated metformin: Women with PCOS who initiated metformin at least 3 months prior to enrollment who have completed a 6-10 day course of progesterone

INTERVENTIONS:
Drug: Endometrin (progesterone 100mg vaginal inserts) — once a day, 6-8 days as specified (prior to each EMBx)
  Groups: A; B
Drug: Metformin — per clinical care guidelines
  Groups: A

SUMMARY:
The investigators aim is to conduct a prospective un-blinded pilot study of premenopausal women diagnosed with Polycystic Ovarian Syndrome (PCOS), defined using criteria developed at the 1990 NICHD conference on PCOS, undergoing treatment for ovulation induction with Metformin. We propose that improving insulin sensitivity with use of Metformin in women diagnosed with PCOS has facilitatory influences on the uterine endometrium.

DETAILED DESCRIPTION:
Endometrial assessments are proposed following three month and then nine month treatment with metformin; expression of specified markers at respective time points will be compared to baseline.

Visit 1: Screening

* Signed informed consent
* Comprehensive history intake
* Physical exam: Vital signs, height, weight, waist circumferences, waist : hip ratio
* Urine pregnancy test
* Subjects provided with a 10 day supply of vaginal progesterone and EMBx will be scheduled between days 6-8 of progesterone use.

Visit 2: Baseline

* Urine pregnancy test
* Endometrium thickness will be measured via transvaginal ultrasound
* EMBx: sample of endometrial tissue will be sent for histopathology to rule out endometrial hyperplasia or cancer
* 20cc blood
* Metformin prescription and dispensing will be as per clinical care.
* Women will be advised to use barrier method of contraception (ie; condoms, contraceptive jellies or foam, sponge, diaphragm, or cervical cap) for the duration of the study.

Visits 3 and 5 (Weeks 8-10 and 30-34, respectively)

* Urine pregnancy test
* A 10 day course of vaginal progesterone to allow scheduling of EMBx's time points specified under visit 1

Visits 4 and 6 (Weeks 12 ± 1 week and 36 ± 1 week respectively)

- The procedure specified for baseline (Visit 2) will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal between 18-42 years of age
* Diagnosed with PCOS as defined by chronic oligo- or amenorrhea (8 menstrual periods annually); biochemical hyperandrogenemia (elevated total or free testosterone) and /or clinical hyperandrogenism (excessive facial hair &/or acne); exclusion of common medical disorders (normal thyroid function tests and serum prolactin and exclusion of 21-hydroxylase deficiency by a fasting 17-hydroxyprogesterone <200 ng/dl).
* Acceptable health on the basis of interview, medical history, physical examination, and laboratory tests (CBC, SMA20, urinalysis) performed within the past 6 months
* Able to provide signed informed consent
* Able to comply with study requirements
* Willing to delay the start of clinically prescribed metformin treatment

Exclusion Criteria:

* Known diabetics or those with clinically significant and known pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, neoplastic and malignant disease (other than non-melanoma skin cancer)
* Current use of hormonal contraceptives
* Seeking pregnancy; use of fertility drugs within 6 months of study
* Current or recent (within 3 months) use of metformin
* Ingestion of any investigational drug within two months prior to study onset
* Evidence of endometrial hyperplasia or cancer upon baseline EMBx

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women will be recruited from the multi-physician Yale Reproductive Endocrinology clinical practice and Yale Fertility Center. Metformin is a routinely employed therapeutic strategy utilized for managing PCOS by practitioners at YFC. Almost 1/3 of the patients with PCOS are not interested in pursuing fertility in the immediate future and it is these patients who will be offered participation in the trial.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
It is anticipated that endometrial expression of implantation markers will be upregulated by metformin treatment compared to baseline and improved parameters will be identified with longer duration of metformin exposure. endometrium biopsy | baseline
It is anticipated that endometrial expression of implantation markers will be upregulated by metformin treatment compared to baseline and improved parameters will be identified with longer duration of metformin exposure. endometrium biopsy | 3 months
It is anticipated that endometrial expression of implantation markers will be upregulated by metformin treatment compared to baseline and improved parameters will be identified with longer duration of metformin exposure. endometrium biopsy | 9 months

SECONDARY OUTCOMES:
blood draw (20mL) | on day of EMBx
A combination of quantitative real time PCR, immunohistochemistry, and Western Blot techniques will be utilized for studying endometrial markers of receptivity in the endometrial tissue | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lubna Pal, MBBS MRCOG MSc, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital Women's Center, New Haven, Connecticut, United States

REFERENCES:
- See also: MedlinePlus related topics: Polycystic Ovary Disease — http://www.nlm.nih.gov/medlineplus/ency/article/000369.htm
- See also: Drug Information available for: Metformin — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a696005.html